CLINICAL TRIAL: NCT00615940
Title: A Phase 2, Two-arm, Double-blind, Multi-center, Randomized Study of the Combination of Oral WX-671 Plus Capecitabine vs. Capecitabine Monotherapy in First-line Her2-negative Metastatic Breast Cancer
Brief Title: Combination of Oral WX-671 Plus Capecitabine vs. Capecitabine Monotherapy in First-line Her2-negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WX/60-006
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2negative
MeSH Terms: conditions — Breast Neoplasms | interventions — upamostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Capecitabine, 1000 mg/m2, twice daily by mouth, on Days 1 to 14, followed by a 7 day rest in each 21 day cycle given in combination with WX-671 once daily by mouth, Days 1-21 inclusive.
  Interventions: Drug: WX-671
- 2 (Experimental): Capecitabine, 1000 mg/m2, twice daily by mouth, on Days 1 to 14, followed by a 7 day rest in each 21 day cycle given in combination with placebo once daily by mouth, Days 1-21 inclusive.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: WX-671 — capsules taken per os once daily until progression or toxicity
  Arms: 1
Drug: placebo — capsule taken per os once daily until progression or toxicity
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo controlled phase II trial is studying how well capecitabine works when given in combination with WX-671 or when given alone in treating patients receiving first-line therapy for her2negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 18 years
* Patients appropriate for palliative first-line, mono chemotherapy with capecitabine
* Histological or cytological confirmed, non-inflammatory metastatic breast cancer
* Availability of paraffin-embedded tumor tissue from the primary resection or biopsy of a metastatic lesion.
* HER2-negative breast cancer
* Complete staging within 2 weeks prior to randomization (4 weeks for bone scan).
* Radiologically confirmed disease
* ECOG performance status of ≤ 2
* Ability to understand and willingness to voluntarily sign and date a written informed consent form before screening
* Negative pregnancy test (urine or serum) within 3 days before first study drug for women of childbearing potential. Use of effective contraception during the study and for 3 months after stopping study drug treatment.
* Normal organ and marrow function as defined by laboratory parameters (obtained within the screening period) within the following limits:

  * neutrophils >= 1.5 x 109/L;
  * platelets >= 100 x 109/L;
  * hemoglobin >= 9.0 g/dL (5.6 mmol/L).
  * total bilirubin <= 1.5 x upper limit of normal (ULN);
  * aspartate aminotransferase (AST)/ALT <= 2.5 x ULN (< 5.0 x ULN for patients with liver metastases);
  * serum creatinine <= 2 x ULN, or calculated creatinine clearance >45 mL/min according to Cockroft and Gault formula).

Exclusion Criteria:

* Endocrine therapy completed within 2 weeks before the start of treatment (i.e. previous hormone therapy is allowed provided that there is a washout period of 2 weeks).
* Prior chemotherapy or biologic therapy for metastatic disease.
* Major surgery within 4 weeks prior to the start of treatment.
* Other anti-cancer treatment (e.g. hormones) within 2 weeks before the start of treatment.
* Treatment within 12 months with adjuvant 5-FU containing chemotherapy (regarded as indicating 5-FU resistance) and/or prior capecitabine therapy.
* Radiation therapy. Palliative radiation of stable, non-target lesions more than 2 weeks before the start of treatment is allowed, provided patients have recovered from the radiation side-effects.
* History of or radiological evidence of brain metastasis including previously treated, resected or asymptomatic brain lesions or leptomeningeal involvement.
* Active seizure disorder or history of cerebrovascular accident (CVA) or transient ischemic (TI) attack within the past 12 months.
* History of other malignancy within the last 3 years except for surgically cured non-melanoma skin cancer or cervical carcinoma in situ.
* Active cardiac disease e.g. unstable angina, congestive heart failure, myocardial infarction (MI) within the preceding 6 months.
* Any medical condition prohibiting standard imaging procedures
* Pregnant or breast-feeding.
* Any unrelated illness, e.g. active infection requiring parenteral antibiotics, inflammation, medical condition or laboratory abnormalities, which in the judgment of the investigator might significantly affect patients' study participation.
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of either study drug.
* Known hepatitis B/C or HIV (human immunodeficiency virus) infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of progression-free survival (PFS) | disease staging with CT/MRI/bone scans at regular intervals

SECONDARY OUTCOMES:
Secondary endpoints are objective response rate (ORR), overall survival, safety and pharmacokinetics. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lori Goldstein, MD, Principal Investigator — Dept. of Medical Oncology, Division of Medical Science, Fox Chase Cancer Center, 7701 Burholme Avenue, Philadelphia, Pennsylvania 19111, USA; Nadia Harbeck, MD, Principal Investigator — Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Uniklinik Köln
Locations (20):
- United States (3):
  - Montefiore Medical Center Weiler Division Department, New York, New York
  - Universitys Hospital Case Medical Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Belgium (3):
  - AZ Klina, Oncology Department, Brasschaat
  - Institut Jules Bordet Oncologie Médicale, Brussels
  - CHU de Liège, Domaine Universitaire de Sart-Tilman, Oncology Department, Liège
- Brazil (3):
  - Irmandade de Misericórdia da Santa Casa de Porto Alegre, Porto Alegre
  - Instituto Nacional do Câncer - INCA, Rio de Janeiro
  - Instituto Brasileiro de Controle do Câncer - IBCC, São Paulo
- Germany (7):
  - Gemeinschaftspraxis Dr. Brudler, Dr. Heinrich, Dr. Bangerter, Augsburg
  - Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Uniklinik Köln, Cologne
  - Universitätsklinikum Essen, Innere Klinik und Poliklinik (Tumorforschung), Essen
  - Uniklinik Frankfurt, Zentrum der Frauenheilkunde und Geburtshilfe, Frankfurt am Main
  - Universitätsklinikum der Martin-Luther-Universität Halle-Wittenberg, Poliklinik Gynäkologie, Halle
  - Bethesda KH, Mönchengladbach
  - Department of Obstetrics and Gynecology, Technical University, Munich
- Israel (4):
  - Davidof Center, Rabin Medical Center, Department of Oncology, Petah Tikva
  - Kaplan Medical Center, Department of Oncolocy, Rehovot
  - Sheba Medical Center, Department of Oncology, Tel Litwinsky
  - Assaf Harofeh medical center, Department of Oncology, Ẕerifin